CLINICAL TRIAL: NCT02366715
Title: IMLEMENTATION OF High Flow Nasal Cannulae Therapy FOR THE TREATMENT OF BRONCHIOLITIS IN A GENERAL PEDIATRIC WARD - A RETROSPECTIVE AND PROSPECTIVE CLINICAL TRIAL
Brief Title: Treatment Of Bronchiolitis With Heated Humidified High Flow Nasal Cannula - Prospective And Retrospective Research
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0586-14-RMC
Record Dates: First submitted 2014-12-22; First posted 2015-02-19 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HeatedHumidifiedHighFlowNasalCannula (Experimental): Treatment for moderate-severe cases of Bronchiolitis while monitoring medical parameters
  Interventions: Device: HeatedHumidifiedHighFlowNasalCannula

INTERVENTIONS:
Device: HeatedHumidifiedHighFlowNasalCannula — We will enroll children 0-2 years old, diagnosed with Bronchiolitis in our ward (Pediatrics C) during the months of November-March 2014-2016. Children will be evaluated according to a Bronchiolitis Severity Score devised by Wang and Co. [3] which was successfully used in previous research. Children answering criteria for moderate or severe Bronchiolitis according to Wang and Co. will be enrolled pending written consent by both parents.
  Our prediction is to enroll a total of 200 children during the 2 winter seasons during 2014-2016.
  Other Names: AIRVO2

SUMMARY:
Bronchiolitis is an acute lower airway infection caused by a viral infection. It is a major cause of winter admissions to pediatric wards. Accepted therapies include oxygen support and IV fluids, whereas other supportive therapies such as inhalations are of questionable benefit. Moderate to severe cases are a source of distress to patient, parents and medical staff often necessitating Pediatric Intensive Care Unit admission. Heated Humidified High Flow Nasal Cannula (HHHFNC) therapy has been shown lately to improve the work of breathing, oxygen saturation, and CO2 pressure (PCO2) values as well as decrease PICU admissions and intubation rates. We planned a prospective and retrospective study in order to check the feasibility of using HHHFNC in a primary pediatric ward and its effect on clinical well being, respiratory status and PICU admission.

DETAILED DESCRIPTION:
Supportive Care, Single Group Assignment, Open Label, Non-Randomized, Efficacy Study

The research is devised as follows:

Prospective section: We will enroll children 0-2 years old, diagnosed with Bronchiolitis in our ward (Pediatrics C) during the months of November-March 2014-2016. Children will be evaluated according to a Bronchiolitis Severity Score devised by Wang and Co which was successfully used in previous research. Children answering criteria for moderate or severe Bronchiolitis according to Wang and Co. will be enrolled pending written consent by both parents.

Our prediction is to enroll a total of 200 children during the 2 winter seasons during 2014-2016.

Retrospective section: We will examine up to 200 cases of children aged 0-2 years hospitalized due to Bronchiolitis in Pediatrics C during 2014-2016 which were not enrolled in our research (due to lack of consent/unavailable HHHFNC etc.). We will compare clinical data and vital parameters between the groups treated with HHHFNC and those who were not.

ELIGIBILITY:
Inclusion Criteria:

in age interval, diagnosed with Bronchiolitis

Exclusion Criteria:

Chronic heart/lung disease, immunocompromised state

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Bronchiolitis Severity Score grade | during the 20-40 hours of the protocol
  The grade in the Bronchiolitis Severity Score (0-12) reflects a general improvement or deterioration in any of these 5 parameters - oxygen saturation, breath rate, general appearance, degree of dyspnea and lung auscultation result.

SECONDARY OUTCOMES:
CO2 pressure | during the 20-40 hours of the protocol
  (in mmHg) measured by a transcutaneous sensor.
Medical interventions | during the 20-40 hours of the protocol
  Any medication given to the child during the time of the protocol including IV fluids, inhalations, diuretics.
Ability to take in food orally | during the 20-40 hours of the protocol
  Whether the child has been able to feed - yes or no.
Number of Pediatric Intensive Care Unit (PICU) admissions | The whole hospitalization period of the child
  Whether the child needed admission to PICU

CONTACTS AND LOCATIONS:
Overall Officials: Eran Rom, Dr., Principal Investigator — Schneider Children Medical Center of Israel
Locations (1):
- Schneider Medical Center of Israel, Petah Tikva, Israel